CLINICAL TRIAL: NCT04159883
Title: The Effect of Using Smart Phone Application for Enhancing Adherence to Home Exercise Program Among Older Adults With Knee Osteoarthritis in Saudi Arabia
Brief Title: The Effect of Using Smart Phone Application for Enhancing Adherence to Home Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Maryam Mohammed Alasfour, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 437203559
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- app (Experimental): For the App group, we installed the app from the store in their smart phone or tablets, made their account using the same email they use in their smart phone store. the participant was informed if they cannot follow the animated image in the app, they can re-launch the program and start to follow.
  Interventions: Other: strengthening exercise program for lower-extremity muscles (knee extensor and hip abductor muscles); Other: "My Dear Knee" smart phone application
- paper (Active Comparator): For the paper group, the participants were provided with a hard copy of the exercise program; we gave one paper of all nine exercises.
  Interventions: Other: strengthening exercise program for lower-extremity muscles (knee extensor and hip abductor muscles)

INTERVENTIONS:
Other: strengthening exercise program for lower-extremity muscles (knee extensor and hip abductor muscles) — Simple progressive strengthening exercise program for lower-extremity muscles (knee extensor and hip abductor muscles), the program has been evident to be significantly effective in improving self-reported knee pain and function. This program included: 1) Isometric quadriceps contraction, 2) Isotonic quadriceps contraction, 3) Isotonic hamstring contraction, 4) Isotonic quadriceps contraction with resistance band, 5), straight leg raising, 6) Side-lying hip abduction, 7) Partial Squats,
Other: "My Dear Knee" smart phone application — The innovative app has been designed for Android and iPhone Operating System (iOS). The app provides guides with the Arabic language. It designed to be attractive for the older adult and easy to use. the exercises are demonstrated with colorful animated images to make easy to follow by the patients.
  The app supports features such as alerts, monitoring system by the physical therapist and remote follow-up. The app provides automatic recording of exercise adherence, including the time and the number of sessions completed for the week in the physical therapist's account.
  Arms: app

SUMMARY:
Background: Knee osteoarthritis (OA) is a serious condition and requires good adherence to interventions such as exercises to achieve optimal management. The use of smart phone technologies could be such a strategy to enhance adherence to the home exercise program (HEP) thus improve pain, physical function and lower limb strength. The study aimed to examine the effect of using an innovative smart phone app on enhancing the adherence to home exercise programs among female older adults with knee OA in Saudi Arabia and the effectiveness of this HEP which delivered through an app, on pain and physical function. Methodology: 40 females aged 50 years or older with knee OA (20 per study arm) recruited to a randomized control trial that uses a parallel study design. All participants assessed and received an education and a set of a home exercise program for knee OA, Participants randomized into the App arm (experimental group) received their HEP in the smart phone application. Participants randomized to the other arm (control group) received HEP in a paper hand-out. After enrolment, the study outcomes were assessed at week three and week six. The primary outcomes were self-reported adherence, ANPRS, and Ar-WOMAC.

ELIGIBILITY:
Inclusion Criteria:

* Female older adults aged 50 and above.
* Diagnosed with unilateral or bilateral chronic knee OA (diagnosed ≥ six months).
* Mild to moderate pain intensity (score ≤ 7 on the Arabic Numeric Pain Rating Scale).
* Ambulate independently.
* Literate, familiar to use smart mobile phone or tablet.
* No previous exercising within the last six months.

Exclusion Criteria:

* Comorbidities that affect their health and wellness (neurological conditions, unstable cardiopulmonary conditions, mental disorders with score < 24 on Mini-Mental State Examination)
* Waiting for surgical intervention.
* Recent trauma (fall/ accident).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The self-reported adherence | 6 weeks
  Adherence rate obtained as a percentage of the exercise done out of the total number of prescribed exercises. The self-reported adherence is a self-report, all the participants received an exercise log and asked to check on the date of the completed exercise. To calculate adherence, the total number of done exercises for each participant was divided by 84 and 182, which were the total number of prescribed exercises for the 3rd and 6th week period respectively.
The Arabic Numeric Pain Rating Scale (ANPRS) | Change from baseline pain score at 6 weeks
  Pain intensity over the previous week evaluated with The Arabic Numeric Pain Rating Scale (ANPRS) which is a reliable and valid scale for assessing pain in knee osteoarthritis. It is a 0 to 10 numerical rating scale in which "0" indicates "no pain" and "10" indicates "worst pain".
The Arabic version of the reduced WOMAC index (ArWOMAC)- Function sub-scale | Change from baseline functional score at 6 weeks
  Used to assess the physical function. It is reliable and valid measure for assessing the severity of knee OA in term of pain and physical function. The reduced ArWOMAC has two subscales and twelve elements in total, the pain subscale includes five elements and the physical function subscale includes seven elements. Likert-scale is applied where the response of each element comes with five levels showing varying intensity degrees that range from 0 to 4, where four is assigned for "extreme" and 0 assigned for "none". The analysis entails collecting and summing up the scores for elements in both subscales to get the total scores (for pain 0-20, for function the scores are 0-28

SECONDARY OUTCOMES:
The Five-Times Sit-To-Stand Test (FTSST) | Change from baseline strength score at 6 weeks
  To evaluate lower-limb muscle strength, the five-times sit-to-stand test used. It is a part of the Short Physical Performance Battery instrument; it is simple, fast, inexpensive and reproducible. It is valid (115) and has excellent test-retest reliability for older adults in general and osteoarthritic older adults. The test utilized an armless chair; the seat rises 46 cm above the ground. The participant starts out by sitting on the chair with arms crossed over the chest. Awarding points is a function of the required time to complete the test. The contributor takes 4 points for the time, not exceeding 11.19 seconds; 3 points when the consumed time is greater than 11.20 and less than 13.69 seconds; two points when the required time ranges from 13.70 and 16.69 seconds; one point if the consumed time is greater than 16.7 seconds; 0 points if the participant cannot complete the test or need more than 60 seconds to finish it.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Almarwani, PhD, Study Director — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with the principal investigator (Mrs. Maryam Alasfour) and sub-investigator (Dr. Maha Almarwani) due to confidentiality issues

REFERENCES:
- [Derived] Alasfour M, Almarwani M. The effect of innovative smartphone application on adherence to a home-based exercise programs for female older adults with knee osteoarthritis in Saudi Arabia: a randomized controlled trial. Disabil Rehabil. 2022 Jun;44(11):2420-2427. doi: 10.1080/09638288.2020.1836268. Epub 2020 Oct 25. PMID 33103499